CLINICAL TRIAL: NCT05430646
Title: Evaluation of Curative Effect of Covered Metal Ureteral Stents in the Endoscopic Treatment of Benign Short Ureteral Stricture: a Prospective Controlled Study
Brief Title: Covered Metal Ureteral Stents in the Treatment of Benign Short Ureteral Stricture
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Huhao, Professor, Peking University People's Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: URO-03
Record Dates: First submitted 2022-06-13; First posted 2022-06-24 (Actual); Last update posted 2022-06-24 (Actual); Status verified 2022-06

CONDITIONS: Ureteral Stenosis
Keywords: ureteral stricture; ureteral stent; curative effect

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CMUS group (Experimental): Balloon dilatation and CMUS insertion were performed in this group.
  Interventions: Device: Covered metal ureteral stents
- Tandem DJ stent group (Active Comparator): Balloon dilatation and Tandem DJ stent insertion were performed in this group.
  Interventions: Device: Tandem DJ stents

INTERVENTIONS:
Device: Covered metal ureteral stents — The CMUS is a fully covered, self-expanding, large caliber metal stent. The stent is made of super-elastic nickel-titanium alloy, which maintain lumen patency via providing long-term direct wall support.
  Arms: CMUS group
Device: Tandem DJ stents — Tandem DJ stents represents for two stents side-by-side, which improves the urine flow by better withstanding the compressive tumoral forces and allowing urine to flow between the stents.
  Arms: Tandem DJ stent group

SUMMARY:
BSUS patients were prospectively enrolled in this study, and non-randomly treated with "balloon dilation +CMUS" and "balloon dilation + tandem DJ stent". Perioperative data of the patients were recorded to compare their efficacy and complications, and the ureteral stent symptom questionnaire was used to compare their impact on patients' quality of life. CMUS and tandem DJ stents were removed after ≥3 months of indwelling. After the removal of stents, the patients' serum creatinine and renal pelvis width were followed up to compare their curative effect on BSUS.

DETAILED DESCRIPTION:
The ureteral stricture is caused by various benign and malignant reasons, and then appears hydronephrosis and progressive decline of renal function. Benign short ureteral stenosis (BSUS) especially refers to ureteral stenosis of no more than 2cm in length caused by benign causes such as impacted ureteral stone or endoscopic lithotomy. Currently, BSUS can be treated with laparoscopic or open ureteroplasty, endoscopic balloon dilation or ureterotomy, ureteral stents insertion, or nephrostomy. Since its introduction, covered metal ureteral stent (CMUS) can be used to treat various types of ureteral stricture, achieving a long-term patency rate of more than 80% for BSUS and even curing some patients. It also has fewer complications than a double-J stent (DJ stent). However, there is still a lack of comparative studies on the therapeutic effect and complications of the two treatment methods, namely CMUS after balloon dilation and tandem DJ stent, for BSUS, especially the evaluation of the curative effect of BSUS. Therefore, BSUS patients were prospectively enrolled in this study, and non-randomly treated with "balloon dilation +CMUS" and "balloon dilation + tandem DJ stent". Perioperative data of the patients were recorded to compare their efficacy and complications, and the ureteral stent symptom questionnaire was used to compare their impact on patients' quality of life. CMUS and tandem DJ stents were removed after ≥3 months of indwelling. After the removal of stents, the patients' serum creatinine and renal pelvis width were followed up to compare their curative effect on BSUS.

ELIGIBILITY:
Inclusion Criteria:

* BSUS patients from January 2023 to January 2024 in Peking University People's Hospital, no gender limitation, aged from 18 to 80, Benign ureteral stricture with definite reason (ureteropelvic junction obstruction, ischemic ureter stenosis caused by surgical separation, ureter partial excision anastomosis stricture after operation, ureteral stricture caused by ureteral endoscope surgery, ureteral stenosis caused by impacted ureteral calculi, ureteral anastomotic stricture after urinary flow diversion, ureteral anastomotic stricture after kidney transplantation, retroperitoneal fibrosis, ureteral stricture caused by trauma, idiopathic ureteral stricture), patients can tolerate anesthesia and surgery and obtain informed consent.

Exclusion Criteria:

* Patients with hypertonic neurogenic bladder, severe bladder outlet obstruction or bladder capacity less than 50ml, combined with sepsis, incomplete clinical data, failed stent implantation, insufficient indwelling time (< 3 months), postoperative loss of follow-up.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Postoperative Serum Creatinine (SCr) | Postoperative 3-month
  It represents for the renal function change after ureteral stent insertion.
Serum Creatinine (SCr) after stent removal | Three-month after stent removal
  It represents for the curative effect of balloon dilatation and ureteral stent.
Postoperative Renal pelvic width (RPW) | Postoperative 3-month
  It represents for the change of hydronephrosis after ureteral stent insertion.
Renal pelvic width (RPW) after stent removal | Three-month after stent removal
  It represents for the curative effect of balloon dilatation and ureteral stent.
Ureteral stent symptom questionnaire (USSQ) | Postoperative 3-month
  USSQ represents for the quality of life of patients with ureteral stents.

SECONDARY OUTCOMES:
Complications | Postoperative 3-month
  Ureteral stent related complications

IPD SHARING:
Plan to Share IPD: No